CLINICAL TRIAL: NCT06219954
Title: Prevention of Pressure Wound Development With Infrared Thermal Camera
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Arzu İLÇE, Professor, Abant Izzet Baysal University
Other Study IDs: AIBÜ-SBF-BD-01; Büşra Demir (Other: AIBÜ)
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pressure Ulcer
Keywords: pressure wound; braden scale; infrared thermography; thermal image; infrared thermal camera
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pressure wound (PW) is generally defined as localized damage to the skin and subcutaneous soft tissue on a bone protrusion or caused by medical devices. Although it is a preventable complication and one of the quality indicators for healthcare institutions, the prevalence of PW is high.Up to 95% of pressure wounds are preventable, but pressure wounds are only detected when sores become visible. Infrared thermography is used in the physiological and anatomical assessment of skin and subcutaneous tissue abnormalities and in detecting pressure injuries by measuring temperature changes caused by circulatory problems.The aim of the researchers is to compare the development of PW in patients admitted to intensive care by imaging the skin temperature in pressure areas using the traditional method and an infrared camera.

DETAILED DESCRIPTION:
Pressure wound (PW); It is localized skin and/or subcutaneous tissue damage, usually occurring on bony prominences, caused by pressure alone or by a combination of shear and pressure.PW is an important source of infection that increases the mortality and morbidity rates of patients, causes an increase in health care costs, causes patients to feel more pain and prolongs the duration of hospital stay, negatively affects the quality of life and causes physical, social and psychological problems, and is an important source of infection, septicemia, It is a global health problem that causes complications such as osteomyelitis and has begun to be accepted as a quality indicator of nursing care. PW, although the risk factors that cause pressure sores are known, there are evidence-level guidelines for preventing pressure ulcers, treatment methods are known, and technological and scientific developments are made, it still appears as a current and serious health problem today.Considering the results of international studies, it has been shown that the prevalence of pressure wounds varies between 7.2-11.6%, the incidence rates vary between 1.9-54.8%, and if precautions are not taken, pressure sores may develop in approximately 87% of patients hospitalized for a long time.Up to 95% of pressure wounds are preventable, but pressure wounds are difficult to detect at an early stage as they can only be detected when the sores become visible.This is because the metabolic demand of the skin is much lower than that of the muscles, the muscles need more oxygen and are more susceptible to ischemia than the skin and surrounding fatty tissue. In this case, the lesions develop in the deep muscle tissue and gradually reach the skin and become visible.Studies have shown that inflammatory and apoptotic/necrotic changes in the epidermal and dermal layers of the skin occur 3-10 days before surface changes.Therefore, a pressure wound in the early stages is difficult to distinguish visually from healthy tissue that responds normally to pressure-inducing factors. Studies have reported that a period of 1 to 7 days must pass from the moment an injury occurs to the tissue for it to appear visually.Risk factors leading to pressure wounds; It can be detected in advance using traditional methods such as visual assessment and the Braden Risk Scale, but these methods are affected by skin color and only 20-40% of pressure wounds can be detected.Infrared thermal camera is a temperature measurement technique that visualizes body thermal energy produced by cellular metabolism and blood circulation in the human body.In body parts where blood flow is impaired, temperature losses occur due to the slowdown of cellular metabolism. Accordingly, when blood flow in the body increases or decreases, there is an increase or decrease in thermal energy measured by an infrared thermal camera. Thus, the infrared thermal camera can be used for physiological and anatomical evaluation of abnormalities in the skin and subcutaneous tissue. The aim of the researchers is to disrupt the basic wound change by imaging the skin temperature under pressure conditions admitted to intensive care with the traditional method and a split camera. New evaluation tools are needed to detect the distribution and pressure sores in the early stages.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving treatment in intensive care
* Patients aged 18 and over
* Patients with Braden score less than 18 points
* Patients who are not transferred from another intensive care unit
* Patients who can tolerate supine, prone and right/left lateral position changes and turns

Exclusion Criteria:

* Patients with previous acute or chronic skin damage or burns in the observation area
* Patients with Braden score over 18 points
* Patients with full-thickness pressure sores
* Patients with protective dressings on the skin or undergoing hot and cold therapy that may affect the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the research will consist of patients who meet the inclusion criteria in the 3-level intensive care clinics of Bolu İzzet Baysal State Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
Braden Risk Assessment Scale | up to 10 days
  The Braden Scale has 6 subdomains. Sensory perception, mobility, moisture, nutrition and activity from 1 to 4; It is scored as 1 being the worst and 4 being the best. Friction is evaluated on 3 different scores, 1 being the worst and 3 being the best. A score between 6-23 is obtained by calculating a total of 6 different categories.
Body/Pressure Zones Temperature Form Measured by Infrared Thermography | up to 10 days
  Measurements will be made of the reference region centered on T1, one of the regions where the risk of pressure injury is considered to be high. In addition, in order to eliminate the effects of endogenous and/or exogenous factors, the distal part, which is at least 10-15 cm away from the areas to be measured, that is, the T2-centered reference region, which is considered the least risky, will be measured with infrared thermography. The temperature difference (ΔT) between these two regions will be calculated (ΔT = T1-T2). When applying the infrared thermal camera to the patient, measurements will be made from a distance of 30 cm at a 90-degree angle after the curtains in the area where the patient lies, ensuring privacy, and the bed borders are removed and safety precautions are taken to prevent the patient from falling.

CONTACTS AND LOCATIONS:
Locations (1):
- İzzet Baysal Devlet Hastanesi, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No